CLINICAL TRIAL: NCT05604131
Title: Cardiac MRI-guided Deferiprone Therapy for Acute Myocardial Infarction Patients
Acronym: MIRON-DFP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rohan Dharmakumar (Other)
Responsible Party: Sponsor-Investigator, Rohan Dharmakumar, Executive Director, Krannert Cardiovascular Research Center, Indiana University School of Medicine
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13487
Record Dates: First submitted 2022-10-07; First posted 2022-11-03 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Acute Myocardial Infarction Type 1
Keywords: Acute Myocardial Infarction; Intramyocardial Hemorrhage; Deferiprone
MeSH Terms: interventions — Deferiprone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Hemorrhagic Myocardial Infarction - Deferiprone (Active Comparator): Enrolled patients with CMR confirmed presence of intramyocardial hemorrhage
  Interventions: Drug: Deferiprone Tablets
- Non-hemorrhagic Myocardial Infarction - Deferiprone (Active Comparator): Enrolled patients with CMR confirmed absence of intramyocardial hemorrhage
  Interventions: Drug: Deferiprone Tablets
- Hemorrhagic Myocardial Infarction - Placebo (Placebo Comparator): Enrolled patients with CMR confirmed presence of intramyocardial hemorrhage
  Interventions: Drug: Placebo
- Non-hemorrhagic Myocardial Infarction - Placebo (Placebo Comparator): Enrolled patients with CMR confirmed absence of intramyocardial hemorrhage
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Deferiprone Tablets — Deferiprone tablets are the active medication for the active arm of the study groups. Randomization will be done by investigational drug services pharmacist and intervention will be double-blinded to investigators and patients.
  Arms: Hemorrhagic Myocardial Infarction - Deferiprone; Non-hemorrhagic Myocardial Infarction - Deferiprone
Drug: Placebo — Deferiprone placebo is the non-medicated formulation for a control arm of the study groups.
  Arms: Hemorrhagic Myocardial Infarction - Placebo; Non-hemorrhagic Myocardial Infarction - Placebo

SUMMARY:
The objective of this randomized, controlled pilot study is to determine the efficacy of Deferiprone to reduce the amount of free iron inside the hemorrhagic zone of myocardial infarction among hemorrhagic myocardial infarction patients.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥ 18 years
2. Index Anterior wall STEMI
3. Emergency coronary angiogram with primary PCI

Exclusion Criteria

1. Prior history of MI / PCI / coronary artery bypass graft (CABG) within previous 1 year
2. Patients with previous history of left ventricular ejection fraction (LVEF) < 40%
3. Use of investigational drugs or devices 30 days prior to randomization
4. Known allergy or contra-indication to gadolinium/contrast agents
5. eGFR < 30 ml/kg/min
6. Any contraindication against cardiac MRI (such as metal implants)
7. Women who are pregnant or breastfeeding. Women of reproductive potential must have a negative pregnancy test prior to randomization
8. Body weight > 140 kg (or 309 lbs.)
9. Absolute neutrophil count - ANC < 1.5 k/cumm
10. History of Chronic Liver Disease
11. Elevated hepatic enzymes (BOTH ALT and AST) > 2 times of upper normal limit
12. Patients with iron storage disease (hemochromatosis, thalassemia) or who are already treated with iron chelators
13. Any clinically significant abnormality identified prior to randomization that in the judgment of the Sponsor-Investigator or Delegate would preclude safe completion of the study or confound the anticipated benefit of deferiprone.
14. Life expectancy of less than 1 year due to non-cardiac pathology

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-11-08 (Actual); Primary Completion 2029-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Treatment Efficacy | 6 months
  Percentage reduction of hemorrhagic zone iron content by cardiac magnetic resonance at 6 months relative to baseline

SECONDARY OUTCOMES:
Treatment Effect: Clinical Outcomes of Acute Heart Failure | 6 months
  The proportion of subjects who experience an acute heart failure event
Treatment Effect: Clinical Outcomes of Non-Fatal Cardiovascular morbidity | 6 months
  The proportion of subjects who experience other non-fatal cardiovascular morbidity such as recurrent myocardial infarction, ventricular arrhythmia and CVA
Safety and Tolerability - Rate of Discontinuation | 6 months
  Rate of discontinuation of therapy due to side effects
Safety and Tolerability - Severe Side Effects | 6 months
  Rate of severe side effects requiring hospitalization, extension of length-of-stay.
Safety and Tolerability - Reversibility of Side Effects without Treatment | 6 months
  Percentage of Reversible of Side Effects without treatment

OTHER OUTCOMES:
Treatment Effect: Fat Infiltration | 6 months
  Percentage difference of fat infiltration within the hemorrhagic myocardial infarction arms at 6 months between deferiprone and placebo groups

CONTACTS AND LOCATIONS:
Overall Officials: Rohan Dharmakumar, PhD, Principal Investigator — Krannert Cardiovascular Research Center; Keyur P Vora, MD FACP FACC, Principal Investigator — Krannert Cardiovascular Research Center
Locations (1):
- Krannert Cardiovascular Research Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kali A, Kumar A, Cokic I, Tang RL, Tsaftaris SA, Friedrich MG, Dharmakumar R. Chronic manifestation of postreperfusion intramyocardial hemorrhage as regional iron deposition: a cardiovascular magnetic resonance study with ex vivo validation. Circ Cardiovasc Imaging. 2013 Mar 1;6(2):218-28. doi: 10.1161/CIRCIMAGING.112.000133. Epub 2013 Feb 12. PMID 23403335
- [Background] Kali A, Cokic I, Tang R, Dohnalkova A, Kovarik L, Yang HJ, Kumar A, Prato FS, Wood JC, Underhill D, Marban E, Dharmakumar R. Persistent Microvascular Obstruction After Myocardial Infarction Culminates in the Confluence of Ferric Iron Oxide Crystals, Proinflammatory Burden, and Adverse Remodeling. Circ Cardiovasc Imaging. 2016 Nov;9(11):e004996. doi: 10.1161/CIRCIMAGING.115.004996. PMID 27903536
- [Background] Wang G, Yang HJ, Kali A, Cokic I, Tang R, Xie G, Yang Q, Francis J, Li S, Dharmakumar R. Influence of Myocardial Hemorrhage on Staging of Reperfused Myocardial Infarctions With T2 Cardiac Magnetic Resonance Imaging: Insights Into the Dependence on Infarction Type With Ex Vivo Validation. JACC Cardiovasc Imaging. 2019 Apr;12(4):693-703. doi: 10.1016/j.jcmg.2018.01.018. Epub 2018 Apr 18. PMID 29680356
- [Background] Liu T, Howarth AG, Chen Y, Nair AR, Yang HJ, Ren D, Tang R, Sykes J, Kovacs MS, Dey D, Slomka P, Wood JC, Finney R, Zeng M, Prato FS, Francis J, Berman DS, Shah PK, Kumar A, Dharmakumar R. Intramyocardial Hemorrhage and the "Wave Front" of Reperfusion Injury Compromising Myocardial Salvage. J Am Coll Cardiol. 2022 Jan 4;79(1):35-48. doi: 10.1016/j.jacc.2021.10.034. PMID 34991787
- [Background] Dharmakumar R. "Rusty Hearts": Is It Time to Rethink Iron Chelation Therapies in Post-Myocardial-Infarction Setting? Circ Cardiovasc Imaging. 2016 Oct;9(10):e005541. doi: 10.1161/CIRCIMAGING.116.005541. No abstract available. PMID 27894072
- [Background] Dharmakumar R. Colors of Myocardial Infarction: Can They Predict the Future? Circ Cardiovasc Imaging. 2017 Dec;10(12):e007291. doi: 10.1161/CIRCIMAGING.117.007291. No abstract available. PMID 29242241
- [Background] Dharmakumar R, Nair AR, Kumar A, Francis J. Myocardial Infarction and the Fine Balance of Iron. JACC Basic Transl Sci. 2021 Jul 26;6(7):581-583. doi: 10.1016/j.jacbts.2021.06.004. eCollection 2021 Jul. PMID 34368506
- [Background] Guan X, Chen Y, Yang HJ, Zhang X, Ren D, Sykes J, Butler J, Han H, Zeng M, Prato FS, Dharmakumar R. Assessment of intramyocardial hemorrhage with dark-blood T2*-weighted cardiovascular magnetic resonance. J Cardiovasc Magn Reson. 2021 Jul 15;23(1):88. doi: 10.1186/s12968-021-00787-4. PMID 34261494
- [Background] Chen Y, Ren D, Guan X, Yang HJ, Liu T, Tang R, Ho H, Jin H, Zeng M, Dharmakumar R. Quantification of myocardial hemorrhage using T2* cardiovascular magnetic resonance at 1.5T with ex-vivo validation. J Cardiovasc Magn Reson. 2021 Sep 30;23(1):104. doi: 10.1186/s12968-021-00779-4. PMID 34587984
- [Background] Kali A, Tang RL, Kumar A, Min JK, Dharmakumar R. Detection of acute reperfusion myocardial hemorrhage with cardiac MR imaging: T2 versus T2. Radiology. 2013 Nov;269(2):387-95. doi: 10.1148/radiology.13122397. Epub 2013 Jul 11. PMID 23847253
- [Background] Cokic I, Kali A, Yang HJ, Yee R, Tang R, Tighiouart M, Wang X, Jackman WS, Chugh SS, White JA, Dharmakumar R. Iron-Sensitive Cardiac Magnetic Resonance Imaging for Prediction of Ventricular Arrhythmia Risk in Patients With Chronic Myocardial Infarction: Early Evidence. Circ Cardiovasc Imaging. 2015 Aug;8(8):10.1161/CIRCIMAGING.115.003642 e003642. doi: 10.1161/CIRCIMAGING.115.003642. PMID 26259581
- [Background] Cokic I, Kali A, Wang X, Yang HJ, Tang RL, Thajudeen A, Shehata M, Amorn AM, Liu E, Stewart B, Bennett N, Harlev D, Tsaftaris SA, Jackman WM, Chugh SS, Dharmakumar R. Iron deposition following chronic myocardial infarction as a substrate for cardiac electrical anomalies: initial findings in a canine model. PLoS One. 2013 Sep 16;8(9):e73193. doi: 10.1371/journal.pone.0073193. eCollection 2013. PMID 24066038
- [Background] Nair AR, Johnson EA, Yang HJ, Cokic I, Francis J, Dharmakumar R. Reperfused hemorrhagic myocardial infarction in rats. PLoS One. 2020 Dec 2;15(12):e0243207. doi: 10.1371/journal.pone.0243207. eCollection 2020. PMID 33264359
- See also: CARDIO-THERANOSTICS is developing diagnostics and therapeutics for hemorrhagic myocardial infarction — https://www.cardio-theranostics.com/